CLINICAL TRIAL: NCT04760015
Title: Characteristics of Patients With Disruptive Vocalizations Residing in Nursing Homes Supported by the Mobile Gerontopsychiatry Team : Retrospective Study
Brief Title: Characteristics of Patients With Dementia Who Are Screaming in Nursing Homes
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0089
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Dementia
Keywords: Dementia disease; Disruptives vocalizations; agitation; cries; profil; characteristics
MeSH Terms: conditions — Dementia; Psychomotor Agitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with dementia develop behavioral problems over time. Among these, the investigators object screams or cries or disruptives vocalizations. Their cause is multifactorial and their management difficult in nursing homes. Often this patients are polymedicated, sedated or/and isolated.

Many scientific studies are interested in drug and non-drug treatments. In this study, the investigators are looking for a profile for disruptives vocalizations's patients. Thus, the investigators will study the global profile of demented patients residing in EHPAD to determine if there are any similarities between them.

ELIGIBILITY:
Inclusion criteria:

* aged 75 years old and more
* living in nursing homes
* dementia
* agitation and disruptives vocalizations
* twice and more interventions by the Mobile Gerontopsychiatry Team

Exclusion criteria:

- no follow-up after team intervention

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Residents in nursing homes, aged 75 years old and more. They have dementia with agitation, including diruptives vocalizations.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Describe the profile of demented patients | 2 years
  Describe the profile of demented patients with disruptives vocalizations in EHPAD aged 75 and over, for whom an intervention of the Mobile Gerontopsychiatry Team (MGT) is requested.
  Determining the profile of the screaming residents in nursing home : age, sex, type of dementia, severity of dementia (MMSE score), co-morbidities, current treatments, sensory impairments, autonomy, environment (visits, outside workers, activities in the EHPAD, paramedical interventions, …), NPI-ES, psychological state (GDS).

SECONDARY OUTCOMES:
Efficiency of MGT's intervention on screams | 2 years
  Evaluate the effectiveness of the MGT's intervention on cries (increase, decrease, stop, lack of effectiveness).
Determination of predictive factors for MGT's effectiveness. | 2 years
  Determine what are the predictive factors of the effectiveness of the intervention of the MGT (time to call after onset of cries, characteristics of the patient and characteristics of the institution).
Determination if the delay between the symptom's beginning and intervention can influence their effectiveness. | 2 years
  Determine if the delay between the onset of screaming and the intervention of the MGT has an impact on the patient's mortality.
Determination if disruptives vocalizations could be a dementia premorbid symptom. | 2 years
  Determine whether screaming is a pre-morbid clinical sign by studying the time interval between the onset of screaming and the patient's death.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Suzanne Leglise, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC